CLINICAL TRIAL: NCT05945342
Title: Research and Application of Key Technologies for Early Identification, Risk Warning and Comprehensive Intervention of Adolescent Depression
Brief Title: Development and Application of Comprehensive Intervention Techniques for Adolescent Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT2023510
Record Dates: First submitted 2023-05-05; First posted 2023-07-14 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Depressive Disorder; Adolescent
MeSH Terms: conditions — Depressive Disorder | interventions — Escitalopram; Interpersonal Psychotherapy; Psychotherapy; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Simple Medication (Active Comparator): Escitalopram alone treatment
  Interventions: Drug: Escitalopram
- Simple Psychotherapy (Active Comparator): Simple interpersonal psychotherapy group
  Interventions: Other: Interpersonal Psychotherapy for Adolescent
- Medication combined with psychotherapy (Experimental): Medication combined with interpersonal psychotherapy
  Interventions: Other: Escitalopram combined with psychotherapy
- Medication combined with physical therapy group (Experimental): Medication combined with robotic navigational repetitive transcranial magnetic stimulation
  Interventions: Other: Escitalopram combined with rTMS
- Medication combined with sham physical therapy group (Sham Comparator): Medication combined with sham robotic navigational repetitive transcranial magnetic stimulation
  Interventions: Drug: Escitalopram combined with sham rTMS

INTERVENTIONS:
Drug: Escitalopram — The US Food and Drug Administration(FDA) has only approved fluoxetine and escitalopram for the treatment of adolescent depression
  Arms: Simple Medication
Other: Interpersonal Psychotherapy for Adolescent — Interpersonal Psychotherapy for Adolescent(IPT-A), A modified version of interpersonal psychotherapy, is shorter than the standard therapy duration (12-16 sessions), with a total of eight sessions, retaining the structure of the standard IPT but employing a series of strategies to extract the most important components to speed up the time process.
  Arms: Simple Psychotherapy
Other: Escitalopram combined with psychotherapy — The subjects received adolescent interpersonal psychotherapy for adolescent(IPT-A) while taking medication
  Arms: Medication combined with psychotherapy
Other: Escitalopram combined with rTMS — The subjects received Robotic navigational repetitive transcranial magnetic stimulation while taking medication
  Arms: Medication combined with physical therapy group
Drug: Escitalopram combined with sham rTMS — The subjects received sham Robotic navigational repetitive transcranial magnetic stimulation while taking medication
  Arms: Medication combined with sham physical therapy group

SUMMARY:
In order to realize the early identification, risk warning and comprehensive intervention of adolescent depression, this project carried out research on the diagnosis platform of adolescent depression, the construction of suicide risk warning and evaluation system, the development of interpersonal psychotherapy technology (IPT-A), and the rapid intervention technology of robotic navigation repetitive transcranial magnetic stimulation (rTMS). Through the extraction of psychological, peripheral and central biological characteristics of adolescent depression and the establishment of a diagnostic platform, combined with artificial neural network to achieve efficient and accurate identification of high risk of suicide population. Antidepressant drugs combined with psychotherapy and antidepressant drugs combined with rTMS physical therapy were used to improve the clinical effective rate and recovery rate. Finally, a comprehensive prevention and control technology suitable for hospitals, schools and families to participate in.

DETAILED DESCRIPTION:
1. The interaction of symptoms, psychological indicators (including environmental risk factors and neuropsychology), peripheral biology (peripheral neuroimmunity, neurotrophic factors and neuroendocrine related indicators), central biological indicators (neuroimaging, near-infrared functional brain imaging) and brain-derived exosome detection in peripheral blood was constructed based on artificial intelligence technology The network of clinical diagnosis platform, and according to the high and low suicide risk classification of deep learning, the establishment of adolescent depression early identification and suicide risk warning system.
2. To develop a simplified interpersonal psychotherapy technique (IPT-A) for adolescent depression.
3. Research and development of rTMS neuroregulation technology for precise positioning of robot navigation in adolescent depression.
4. Construct comprehensive intervention models and efficacy prediction models for adolescent depression, such as drug combined with psychology and drug combined with physical therapy, and promote and demonstrate the application.

ELIGIBILITY:
Inclusion Criteria:

* Sign a written informed consent to participate in the trial and receive treatment;
* Meet the diagnostic criteria of depression in DSM-5, and have no psychotic characteristics;
* Child Depression Rating Scale-Revised (CRs-R)≥40 points;
* 24 Hamilton Depression Scale (HAMD-24) scores ≥20;
* First or recurrent depressive episode, not received antidepressant drugs and systematic psychotherapy in recent 2 months;
* The Han nationality, right hand

Exclusion Criteria:

* Have other mental disorders, or have a history of other mental disorders, such as attention deficit movement disorder, autism, and developmental retardation;
* Patients with current infections, trauma, autoimmune diseases, other unstable medical conditions, or who are receiving hormone therapy;
* Patients with a history of craniocerebral injury and coma;
* A family history of bipolar disorder, seizures, or epilepsy;
* Those who had substance abuse or dependence within the first three months of enrollment;
* Patients with contraindications for MRI examination such as metal foreign body in the skull or abnormal brain structure found in MRI examination.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Score of Child Depression Rating Scale-Revised | Baseline, 2-week, 4-week, 8-week
  For clinical depression symptom assessment
Score of Beck Scale for Suicide Ideation | Baseline, 2-week, 4-week, 8-week
  For the quantitative assessment of suicidal ideation
Score of Iowa Gambling Task | Baseline, 2-week, 8-week
  The simulation of the real decision situation is a kind of decision making task in the fuzzy situation accompanied by corresponding rewards and punishments
Score of THINC-it test | Baseline, 2-week, 8-week
  The test includes Spotter, Symbol check, Codebreaker, Trails, and the 5-item Depression Cognitive Deficit Questionnaire (PDQ-5-D). It is used to assess working memory, executive function and attention
Hypocretin | Baseline, 2-week, 8-week
  Hypocretin is a neurotransmitter that regulates wakefulness and appetite
Endocannabinoid | Baseline, 2-week, 8-week
  Endocannabinoid play an important role in regulating many functions in the body, including the inflammatory system, immune function, sleep, appetite, digestion, pain receptors, hormones, reproductive function and memory
Neuroimmune-related factors | Baseline, 2-week, 8-week
  Such as IL-lβ、IL-6、TNF-α
Neurotrophic pathway related factors | Baseline, 2-week, 8-week
  Such as BDNF、VGF、TrkB、tPA
Near infrared functional imaging of the brain | Baseline, 2-week, 8-week
  Near infrared functional brain imaging can reflect the activation degree of brain function and functional connectivity of brain by detecting the concentration changes of oxygenated hemoglobin and deoxygenated hemoglobin in the target brain area.
Change in working memory test scores after intervention | Baseline, 2-week, 8-week, 24-week
  The working memory test consists of two parts, which measure the breadth and accuracy of working memory respectively. The breadth of working memory will be tested using the operating span experiment, as the accuracy of working memory will be tested using the Memory Orientation experiment
Change in three component test of executive function scores after intervention | Baseline, 2-week, 8-week, 24-week
  The three component tests of executive function were one-backward test, anti-saccade and shifting test respectively.In the one-backward test, subjects need to memorize letters while counting numbers, scoring them according to the accuracy of the alphabetic memory order; The anti-saccade test asks subjects to react to a flash of arrows (0.5 seconds) by selecting the direction they see on a keyboard；The shifting test asked subjects to select a forward or reverse feedback key depending on where the icon appeared
TMS-Evoked potential | Baseline, 2-week, 8-week
  The integration of transcranial magnetic stimulation (TMS) and electroencephalography (EEG) is a valuable method for directly probing excitability, connectivity and oscillatory dynamics of regions throughout the brain. Offering in depth measurement of cortical reactivity, TMS-EEG allows the evaluation of TMS-evoked components that may act as a marker for cortical excitation and inhibition.
Magnetic Resonance Imaging | Baseline, 2-week, 8-week
  Functional magnetic resonance brain imaging can reflect the functional and metabolic information of neurons before morphological changes

SECONDARY OUTCOMES:
Score of 24-item Hamilton Depression Rating Scale | Baseline, 2-week, 4-week, 8-week
  For clinical depression symptom assessment
Ottawa Self-injury Questionnaire | Baseline, 2-week, 4-week, 8-week
  To evaluate the situation of NSSI among adolescents
Score of Childhood Trauma Questionnaire | Baseline
  Used to assess traumatic experiences in childhood

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided